CLINICAL TRIAL: NCT04081012
Title: N-acetyl Cysteine in Post-reperfusion Pulmonary Injury in Patients With Chronic Thromboembolic Pulmonary Hypertension Undergoing Pulmonary Balloon Angioplasty and Pulmonary Endarterectomy.
Brief Title: N-acetyl Cysteine in Post-reperfusion Pulmonary Injury in Chronic Thromboembolic Pulmonary Hypertension.
Acronym: NAC-PostRep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Maria Elena Soto, MsC and PhD, Clinical Research, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 191110
Record Dates: First submitted 2019-08-16; First posted 2019-09-06 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind clinical trial of the treatment will be the treating physician and radiologist, of parallel groups in patients undergoing EAP and BPA.
Who Masked: Participant, Care Provider, Investigator
Masking Description: It will be through sealed, opaque and numbered envelopes sequentially. The assignment sequence will be done by the pharmacist, the principal investigator will recruit the patients. Researchers and site staff (with the exception of the investigating pharmacologist) will be blinded to the assigned treatment. There will be no circumstances to unmask and reveal the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetyl Cysteine (Experimental): Patients will receive a 4-dose schedule of 600 mg diluted in 50 ml of 0.9% saline intravenously every 12 hours starting 24 hours before endarterectomy or balloon angioplasty.
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): The placebo group will receive a similar volume of normal saline as a placebo at the same time intervals. All study medications will be prepared by the Pharmacology department, which is not involved in patient care; the name of the medication and dose of the original ampule will be erased and also an identification label will be placed with the name, registration number, bed number, date and will be indifferent for groups with the same type of ampoule, with the same type of labeling
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — Patients will receive a 4-dose schedule of 600 mg diluted in 50 ml of 0.9% saline intravenously every 12 hours starting 24 hours before pulmonary endarterectomy or balloon pulmonary angioplasty.
  Other Names: NAC
  Arms: N-acetyl Cysteine
Drug: Placebo — The placebo group will receive a similar volume of normal saline as a placebo at the same time intervals.
  Arms: Placebo

SUMMARY:
This study will evaluate the use of N-acetyl cysteine in post-reperfusion pulmonary injury in patients with chronic thromboembolic pulmonary hypertension undergoing pulmonary balloon angioplasty and pulmonary endarterectomy. Half of the patients will receive N-acetyl cysteine and the other placebo.

DETAILED DESCRIPTION:
For chronic pulmonary embolism thrombus hypertension, the potentially curative treatment is endarterectomy, however in 12 to 60% it does not present surgical susceptibility, so pulmonary balloon angioplasty is the secondary option. In these procedures the complication that occurs most frequently is pulmonary oedema after reperfusion is a frequent complication (17.8-65%), appears between 24-72 hours after the intervention and the diagnosis is made in the presence of infiltrate interstitial in chest radiography or computed tomography of the chest. Initially it was believed that it was difficult due to the increase in perfusion of secondary flow in the territory due to pulmonary vascular dilation, it is now believed that microtraumatism is involved by the guides and balloon used, vascular dysfunction and cytokines and innate immunity and adaptive, complement activation, coagulation cascade activation, apoptosis pathway activation, endothelial dysfunction caused by reperfusion contribute to cell dysfunction.

The use of N-acetyl cysteine for its antioxidant properties, inflammatory response attenuator, reduction of reactive oxygen species (ROS) and that in addition to having already had to reduce the condition of decrease in post-reperfusion ischemia15,16 in other situations is a viable option in the treatment of acute post-reperfusion edema in patients sometimes a pulmonary endarterectomy and balloon pulmonary angioplasty.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are diagnosed with group 4 pulmonary hypertension and are susceptible to pulmonary endarterectomy or balloon angioplasty in patients over 18 years.

Exclusion Criteria:

* Patients who do not accept admission to the trial.
* Presence of arterial hypotension or sepsis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2023-05-21 (Estimated); Study Completion 2023-05-21 (Estimated)

PRIMARY OUTCOMES:
Presence of Post-reperfusion pulmonary injury. | 72 hours
  Chest tomography will be performed using 35 mA, 100 Kv and 6 mm cuts, then the simple thorax (low dose) holding the inspiration in the cephalocaudal direction with 80 mA, 100 Kv, a duration of 2.24 seconds, pitch of 1 and cuts 1 mm Multiplanar reconstructions with Kernel filters B26f, B50f and B70f for mediastinum and lung respectively, at 1 mm cuts. And anteroposterior chest radiographs will be obtained with the same equipment, at the beginning of the study and daily on days 1 to 3.

SECONDARY OUTCOMES:
Concentration of cytokines (pg/ml) | Basal and at 72 hours
  Blood samples for the determination of plasma cytokines will be extracted from the peripheral venous puncture, jugular venous line and / or Swan Ganz catheter in patients undergoing EAP or by pigtail pulmonary artery trunk catheter to patients who are underwent BPA, at the following time points: baseline upon admission to hospital and / or after induction of anesthesia and before the incision (T1), and at 72 hours (T2) after the onset of surgery. All blood samples will receive the same process. immunohistochemistry will be performed for IP-10 (1: 250, ab9807; Abcam, Cambridge, UK), IL-8 (1: 100; ab7747; Abcam), MCP-1 (1: 100, ab73680; Abcam) and IL-6 (1: 100, ab6672; Abcam) will be performed with a 3,39-diaminobenzidine peroxidase substrate from R&D kit Systems (Minneapolis, MN, USA). Specifically for IP-10, IL-8, RANTES, MIG and MCP-1 will be measured by Human Chemokine Kit Cytometric Bead Array (Becton Dickinson, Franklin Lakes, NJ, USA), following the manufacturer's specifications.
Percentaje of Complications (%) | 30 days
  Dead

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elena Soto Lopez, Principal Investigator — Instituto Nacional de Cardiología "Ignacio Chávez"
Locations (1):
- Instituto Nacional Ignacio Chavez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 8 months of study completion.
Access Criteria: Data access request will be reviewed by an internal review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Konstantinides SV, Barco S, Lankeit M, Meyer G. Management of Pulmonary Embolism: An Update. J Am Coll Cardiol. 2016 Mar 1;67(8):976-990. doi: 10.1016/j.jacc.2015.11.061. PMID 26916489
- [Background] Huisman MV, Barco S, Cannegieter SC, Le Gal G, Konstantinides SV, Reitsma PH, Rodger M, Vonk Noordegraaf A, Klok FA. Pulmonary embolism. Nat Rev Dis Primers. 2018 May 17;4:18028. doi: 10.1038/nrdp.2018.28. PMID 29770793
- [Background] Pengo V, Lensing AW, Prins MH, Marchiori A, Davidson BL, Tiozzo F, Albanese P, Biasiolo A, Pegoraro C, Iliceto S, Prandoni P; Thromboembolic Pulmonary Hypertension Study Group. Incidence of chronic thromboembolic pulmonary hypertension after pulmonary embolism. N Engl J Med. 2004 May 27;350(22):2257-64. doi: 10.1056/NEJMoa032274. PMID 15163775
- [Background] Ogawa A, Satoh T, Fukuda T, Sugimura K, Fukumoto Y, Emoto N, Yamada N, Yao A, Ando M, Ogino H, Tanabe N, Tsujino I, Hanaoka M, Minatoya K, Ito H, Matsubara H. Balloon Pulmonary Angioplasty for Chronic Thromboembolic Pulmonary Hypertension: Results of a Multicenter Registry. Circ Cardiovasc Qual Outcomes. 2017 Nov;10(11):e004029. doi: 10.1161/CIRCOUTCOMES.117.004029. PMID 29101270
- [Background] Wilkens H, Lang I, Behr J, Berghaus T, Grohe C, Guth S, Hoeper MM, Kramm T, Kruger U, Langer F, Rosenkranz S, Schafers HJ, Schmidt M, Seyfarth HJ, Wahlers T, Worth H, Mayer E. Chronic thromboembolic pulmonary hypertension (CTEPH): updated Recommendations of the Cologne Consensus Conference 2011. Int J Cardiol. 2011 Dec;154 Suppl 1:S54-60. doi: 10.1016/S0167-5273(11)70493-4. PMID 22221974
- [Background] Laubach VE, Sharma AK. Mechanisms of lung ischemia-reperfusion injury. Curr Opin Organ Transplant. 2016 Jun;21(3):246-52. doi: 10.1097/MOT.0000000000000304. PMID 26945320
- [Background] Zabini D, Heinemann A, Foris V, Nagaraj C, Nierlich P, Balint Z, Kwapiszewska G, Lang IM, Klepetko W, Olschewski H, Olschewski A. Comprehensive analysis of inflammatory markers in chronic thromboembolic pulmonary hypertension patients. Eur Respir J. 2014 Oct;44(4):951-62. doi: 10.1183/09031936.00145013. Epub 2014 Jul 17. PMID 25034560
- [Background] Sun Y, Pu LY, Lu L, Wang XH, Zhang F, Rao JH. N-acetylcysteine attenuates reactive-oxygen-species-mediated endoplasmic reticulum stress during liver ischemia-reperfusion injury. World J Gastroenterol. 2014 Nov 7;20(41):15289-98. doi: 10.3748/wjg.v20.i41.15289. PMID 25386077
- [Background] Geudens N, Wuyts WA, Rega FR, Vanaudenaerde BM, Neyrinck AP, Verleden GM, Lerut TE, Van Raemdonck DE. N-acetyl cysteine attenuates the inflammatory response in warm ischemic pig lungs. J Surg Res. 2008 May 15;146(2):177-83. doi: 10.1016/j.jss.2007.05.018. Epub 2007 Jul 20. PMID 17644109